CLINICAL TRIAL: NCT06907563
Title: Long-term Follow-up to Determine Outcome in Liver Disease (LOVE Study)
Acronym: LOVE
Status: Not yet recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Collaborators: Universitatsmedizin Mainz - 1. Medizinische Klinik (Other); Newcastle University (Other); Barcelona Institute for Global Health (Other); Odense University Hospital (Other); Hospital Clinic of Barcelona (Other); Assistance Publique - Hôpitaux de Paris (Other); University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: LOVE study
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Steatotic Liver Disease; MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); Steatotic Liver Disease of Mixed Origin (MetALD); ALD - Alcoholic Liver Disease
Keywords: MASH; SLD; NITs; MASLD; ALD; MetALD; Metabolism; Liver
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- European SLD Registry: The EU-SLD registry comprises patients from 18 european countries and a study cohort of n=8.984 with most recent cases recruited in the prospective LITMUS cohort study. Now followed up as part of the LOVE Study in the EU-LIVERAIM project.

SUMMARY:
The rational to conduct the LOVE study builds on the lack of available data on outcomes in steatotic liver disease in well characterized patients over a time frame of several years. At current limited data on liver-specific and overall outcome in patients with MASLD, MetALD and ALD are available. Liver histology is the only accepted surrogate to reasonably likely predict outcomes in patients with non-cirrhotic liver disease and is currently used in regulatory trials. To overcome the limitations of liver biopsy and use validated non-invasive tests (NITs) to predict outcomes, the LOVE study will be conducted based on existing cohort studies in well pheno- and genotyped patients and will inform on the relevant outcomes based on baseline and ongoing biomarker assessment. The overarching goal is to qualify a NIT for patient identification and preventive measures in the regulatory context.

ELIGIBILITY:
Inclusion Criteria:

* Previous Informed consent for cohort studies
* > 18 years of age
* Diagnosis of SLD (MASLD, MetALD, ALD)

Exclusion Criteria:

* No consent for previous cohort studies
* < 18 years of age
* No Diagnosis of SLD (MASLD, MetALD, ALD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European SLD register (historically EPOS, LITMUS); 18 european countries.
  https://pubmed.ncbi.nlm.nih.gov/33045403/
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Major-adverse liver outcomes (MALO) | 5 years follow-up time
  Development of cirrhosis. Hepatic decompensation: ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, portal hypertension, varices.
All-cause mortality | 5 years follow-up time
  Death during the follow-up period due to any cause

SECONDARY OUTCOMES:
Health-related quality of life (HRQL) | 5 years
  To measure the impact on the health-related quality of life in patients during the natural history of the disease.
Assess prognostic biomarkers and develop a novel tool to integrate them into a digital tool to predict outcomes | 5 years
Major adverse cardiac events (MACE) | 5 years
Development of relevant clinical outcomes | 5 years
  Incidence of cancer, chronic kidney disease, neurodegenerative disease, dementia, and depression

CONTACTS AND LOCATIONS:
Locations (4):
- Hôpital de la Pitié Salpêtrière, Paris, France
- University Medical Center Saarland, Department of Internal Medicine II, Homburg, Saarland, Germany
- Division of Gastroenterology, Department of Medical Sciences, University of Turin, Turin, Italy
- Translational & Clinical Research Institute Faculty of Medical Sciences, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a plan to make IPD available.